CLINICAL TRIAL: NCT05418634
Title: The Role of Point-of-care EEG in the Pediatric Emergency Department
Brief Title: Point-of-care EEG in the Pediatric Emergency Department
Status: Completed | Type: Observational
Sponsor: University Children's Hospital, Zurich (Other)
Collaborators: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Principal Investigator, Leopold Simma, PEM Attending, University Children's Hospital, Zurich
Other Study IDs: 2022-00842
Record Dates: First submitted 2022-06-09; First posted 2022-06-14 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Status Epilepticus; Non-Convulsive Status Epilepticus; Altered Mental Status
Keywords: pediatric emergency medicine; pediatric neurology; status epliepticus; non-convulsive status epilepticus; altered mental status
MeSH Terms: conditions — Status Epilepticus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Pediatric Emergency Department (PED): PED: Patients presenting with unexplained impaired consciousness or active SE:
  To investigate the role of pocEEG in the PED, we will collect all pocEEG tracings of all children with unexplained impaired consciousness or active SE, for whom written consent has been obtained. We will document the interpretation of the respective pocEEGs by the PEM physician and compare it to the interpretation of the neuropediatrician on call. The research team will also perform a post-hoc analysis.
  Interventions: Other: point of care EEG
- Epilepsy Clinic: CLINIC: Patients with either suspected epilepsy or established diagnosis of epilepsy will be recruited for simultaneous recording of cEEG and pocEEG in the epilepsy outpatient clinic will help define and investigate the limitations of pocEEG.
  Interventions: Other: point of care EEG

INTERVENTIONS:
Other: point of care EEG — For pocEEG, scalp electrodes are applied in five locations.

SUMMARY:
The researchers investigate the use of a simplified electroencephalogram (point-of-care EEG) in the pediatric emergency department for children with impaired consciousness or an ongoing epileptic seizure ("status epilepticus"). In addition, the researchers will compare the simplified EEG with the conventional EEG in the epilepsy outpatient clinic.

DETAILED DESCRIPTION:
Non-traumatic, acute central nervous system (CNS) disorders are amongst the most frequent emergencies in childhood. In Switzerland, CNS disorders are the top ranking presentation of critically ill children. Many pediatric neurological emergencies such as coma, acute encephalopathies with impaired consciousness or agitation, or acute focal deficits, are associated with changes of cortical electrical activity detectable by the electroencephalogram (EEG). Of particular concern are status epilepticus (SE) and non-convulsive status epilepticus (NCSE). Previous studies have shown that an EEG can yield important diagnostic information and aid in decision-making. However, conventional EEG-recordings are resource intensive (time, staff), and hardly available outside of regular working hours. Point-of-care EEG (pocEEG) has proven helpful for evaluating impaired consciousness, detecting NCSE, and monitoring therapy in ongoing SE. In a retrospective cohort study from Japan patients with impaired consciousness were diagnosed with non-convulsive seizures in pocEEG, supporting the view that pocEEG can be applied by ED physicians, even in the absence of a neurologist, and can aid the detection and treatment of non-convulsive seizures. Another study, also from Japan, reported that abnormalities were detected in 20% of patients by using pocEEG in an ED setting. The aims of this study are:

* To prospectively assess the feasibility and utility of pocEEG for NCSE detection in children presenting with impaired consciousness in the PED
* To evaluate the interpretation accuracy of pocEEG by pediatric emergency medicine (PEM) providers after a teaching module.
* To compare pocEEG to the "gold standard" of simultaneously recorded conventional EEG in patients undergoing routine cEEG in the epilepsy outpatient clinics.

ELIGIBILITY:
Inclusion Criteria:

General:

PED:

* Pediatric patients with unexplained impaired consciousness, suspicion of NCSE, active SE presenting to the PED
* Informed consent of patient of parents/persons responsible, if possible, otherwise emergency situation procedure (according to national regulations for research in emergency situations)

CLINIC:

* Informed consent as documented by signature
* Pediatric patients undergoing cEEG in the outpatient epilepsy clinics
* Either suspected/ to rule out epilepsy or established diagnosis of epilepsy

Exclusion Criteria:

PED:

* AMS of known etiology or another diagnosis
* Declined informed consent

CLINIC:

* Failure to provide signed informed consent
* Changes in health condition which might interfere with the EEG recording.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All pediatric patients presenting to the PED or the epilepsy clinic fulfilling the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2022-08-24 (Actual); Primary Completion 2025-08-23 (Actual); Study Completion 2025-08-24 (Actual)

PRIMARY OUTCOMES:
Number of participants diagnosed with SE, NCSE, and encephalitis by pocEEG | Baseline
  All patients with impaired consciousness presenting to the PED will receive a pocEEG. We analyse the number of patients with SE, NCSE, and encephalitis diagnosed by pocEEG
Agreement pocEEG vs. conventional EEG in epilepsy clinic | Baseline
  Agreement of pocEEG and cEEG findings in simultaneous tracings carried out during routine care in the epilepsy clinic.

CONTACTS AND LOCATIONS:
Overall Officials: Georgia Ramantani, MD, PhD, Principal Investigator — University Children's Hospital, Zurich
Locations (1):
- University Children's Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Simma L, Romano F, Schmidt S, Ramantani G, Bolsterli BK. Integrating Neuromonitoring in Pediatric Emergency Medicine: Exploring Two Options for Point-of-Care Electroencephalogram (pocEEG) via Patient Monitors-A Technical Note. J Pers Med. 2023 Sep 20;13(9):1411. doi: 10.3390/jpm13091411. PMID 37763178
- [Background] Simma L, Bauder F, Schmitt-Mechelke T. Feasibility and usefulness of rapid 2-channel-EEG-monitoring (point-of-care EEG) for acute CNS disorders in the paediatric emergency department: an observational study. Emerg Med J. 2021 Dec;38(12):919-922. doi: 10.1136/emermed-2020-209891. Epub 2020 Oct 30. PMID 33127740
- [Background] Nozawa M, Terashima H, Tsuji S, Kubota M. A Simplified Electroencephalogram Monitoring System in the Emergency Room. Pediatr Emerg Care. 2019 Jul;35(7):487-492. doi: 10.1097/PEC.0000000000001033. PMID 28072672
- [Background] Yamaguchi H, Nagase H, Nishiyama M, Tokumoto S, Ishida Y, Tomioka K, Tanaka T, Fujita K, Toyoshima D, Nishimura N, Kurosawa H, Nozu K, Maruyama A, Tanaka R, Iijima K. Nonconvulsive Seizure Detection by Reduced-Lead Electroencephalography in Children with Altered Mental Status in the Emergency Department. J Pediatr. 2019 Apr;207:213-219.e3. doi: 10.1016/j.jpeds.2018.11.019. Epub 2018 Dec 7. PMID 30528574